CLINICAL TRIAL: NCT01768650
Title: Telephone-Delivered Cognitive Behavioral Therapy for Chronic Pain Following Traumatic Brain Injury
Brief Title: Structured Treatment of Pain (STOP) Study
Acronym: STOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeanne Hoffman, Professor, Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 44437
Record Dates: First submitted 2013-01-09; First posted 2013-01-15 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Traumatic Brain Injury; Chronic Pain
Keywords: traumatic brain injury; chronic pain; headache; Veteran
MeSH Terms: conditions — Brain Injuries, Traumatic; Chronic Pain; Headache

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Management #2 (Experimental): Self-Management #2 will consist of eight 60-minute sessions conducted by phone over eight weeks (1 session/week on average). The sessions will cover a variety of topics, including: (1) the definition of chronic pain, (2) the physiological processes underlying chronic pain, (3) common pain-related conditions such as sleep and mood disturbance (including posttraumatic stress disorder, due to its prevalence among Veterans), (4) the potential effects of chronic pain on activity level, (5) communication (including communication with healthcare providers), and (6) the role of social support in managing pain.
  Interventions: Behavioral: Self-Management #2
- Self-Management #1 (Experimental): Self-Management #1 will consist of eight 60-minute sessions conducted by phone over eight weeks. Sessions will include: (1) education about the role of cognitions and pain beliefs (including control) in chronic pain and adjustment; (2) instruction in how to identify negative thinking and cognitive distortions about pain; (3) instruction in thought-stopping and cognitive-restructuring techniques, including challenging negative thoughts and core beliefs about pain; (4) instruction in utilization of positive coping self-statements; (5) relaxation techniques; (6) activity pacing and scheduling; (7) coping with pain flare-ups; and (8) relapse prevention/maintenance of gains. Most sessions will include a brief relaxation exercise introduced over the phone.
  Interventions: Behavioral: Self-Management #1

INTERVENTIONS:
Behavioral: Self-Management #1 — Self-Management #1 will consist of eight 60-minute sessions conducted by phone over eight weeks. Sessions will include: (1) education about the role of cognitions and pain beliefs (including control) in chronic pain and adjustment; (2) instruction in how to identify negative thinking and cognitive distortions about pain; (3) instruction in thought-stopping and cognitive-restructuring techniques, including challenging negative thoughts and core beliefs about pain; (4) instruction in utilization of positive coping self-statements; (5) relaxation techniques; (6) activity pacing and scheduling; (7) coping with pain flare-ups; and (8) relapse prevention/maintenance of gains. Most sessions will include a brief relaxation exercise introduced over the phone.
  Arms: Self-Management #1
Behavioral: Self-Management #2 — Self-Management #2 will consist of eight 60-minute sessions conducted by phone over eight weeks (1 session/week on average). The sessions will cover a variety of topics, including: (1) the definition of chronic pain, (2) the physiological processes underlying chronic pain, (3) common pain-related conditions such as sleep and mood disturbance (including posttraumatic stress disorder, due to its prevalence among Veterans), (4) the potential effects of chronic pain on activity level, (5) communication (including communication with healthcare providers), and (6) the role of social support in managing pain.
  Arms: Self-Management #2

SUMMARY:
This study seeks to compare two different behavioral treatments for pain in Veterans with a history of TBI. Both treatments involve educating the Veteran about pain, discussing the impact of pain, and different ways to manage it in hopes of decreasing pain and its impact on life. These approaches are called "self-management" approaches to pain. Both of these treatments are commonly used in pain clinics to treat pain in persons with back pain, headaches, and other types of chronic pain. The investigators will be delivering both treatments over the telephone to make the treatments accessible to Veterans wherever they live.

DETAILED DESCRIPTION:
People with a history of traumatic brain injury (TBI) often have pain, such as headaches or neck pain as well as pain from other injuries. Effective treatments that teach people how to manage pain have been used to treat chronic pain in the general population. However, it is often hard for people to access these treatments, as since they are usually only offered in person. The investigators are interested in learning if these treatments can be effectively delivered by telephone, and if the treatments are effective for Veterans with a history of TBI. The purpose of this study is to compare two of these treatments to see if they can be delivered by telephone, and see if they can help reduce pain in Veterans with a history of TBI. Both of these methods are called "self-management" approaches to pain management. Both of these treatments are commonly used in pain clinics and have been used to treat pain in persons with TBI. The investigators are interested in comparing these two different approaches to self-management delivered by phone. Additionally, the investigators want to determine if these treatments can help reduce the negative consequences that pain often causes, such as disruption in mood, daily activities, and enjoyment of life.

The sponsor of this study is the Department of Defense. The scientist in charge of this project is at the University of Washington, as are many of the co-investigators and study staff. However, all the people who participate in this study will be Operation Enduring Freedom (OEF)/Operation Iraqi Freedom (OIF)/Operation New Dawn (OND) Veterans recruited from VA Puget Sound Health Care System (VAPSHCS). Dr. Rhonda Williams is the scientist at the VAPSHCS who will oversee the project activities at this site. The investigators enrolled 231 subjects into this study. The study will be funded through September 29, 2017.

Subjects will be asked to participate in the following:

1)Informed Consent 2)6 Six Assessments (including cognitive testing, interviews administered by phone and in person) 3)Participate in a telephone-based 1:1 treatment intervention for pain. Subjects will be randomly assigned (by chance, like flipping a coin) to one of the two treatment interventions.

4)All of the activities included in the study are considered research and would not normally be part of the treatment subjects receive at the VAPSHCS.

Details about the various study activities are included below:

Informed Consent A research staff member will review the details of the study with each subject and answer any questions the subject may have, and see if the subject is interested in participating. Subjects will then print their name, sign and date the study consent form if they are interested in participating.

Assessments There are several assessments required as part of subjects' participation in this study: cognitive tests, a baseline assessment interview, and four "assessment periods". The "assessment periods" are weeks in which the researchers will call subjects four times, each on a different day, to do a brief assessment interview. All of these assessments are described in detail below.

Cognitive Testing Session

The first assessment is a short battery of cognitive tests. These tests will test memory and information processing. These tests will take about 15-20 minutes to complete and need to be completed in person. Subjects can complete them immediately following the consent process today or at a later time. Subjects will be compensated $20 for completing this assessment.

Baseline Assessment Interview A research staff member will interview each subject for 20-30 minutes. Subjects will be asked a number of standard questions such as their age, gender, race, ethnicity, education level, military service, and their pain problem(s). Research staff members will also ask about personal habits and history, including alcohol and drug use, as well as any problems subjects may experience related to stressful military experiences. Subjects will also be asked two questions about whether or not they ever experienced military sexual trauma. These questions will take about 20-30 minutes to answer all together, and can be completed in person after the cognitive testing session, or over the telephone at a later time. Subjects will not be paid to complete this interview.

Medical Record Review

Research staff members will collect some information about subjects from their medical record, including the following:

Level of Service Connection Number of TBI-Related Events Where subjects were located when the TBI-Related Events occurred (e.g., in combat, in the USA) Causes of TBI(s) Severity of TBI(s)

This information will be linked to the data subjects provide while participating in the study. Subjects will not have to do anything other than enroll in the study in order for the researchers to review their medical records.

Four Telephone Assessment Periods Research staff will call subjects to complete four sets of telephone interviews during study participation. The first of these will occur at the beginning of the study. The second will occur about half- way through treatment. The third will occur at the end of treatment, and the fourth will occur about six months after the subject began treatment. Each assessment period will include four telephone calls on different days, all within the same week. Telephone calls may be as brief as 5 minutes, or one of the 4 lasting as long as 30 minutes, depending on how subjects choose to space the assessment questions over the four calls within a given assessment period week. The entire assessment will take about 40-45 minutes to complete, spread over four telephone calls within a week.

During each telephone call, research staff will ask subjects at the minimum to rate their current, average, worst and least pain intensity over the past 24 hours, as well as the frequency and severity of any headaches subjects may have had in the past 24 hours.

In addition, once during each of the four assessment period weeks the research staff will also ask subjects an extra set of questions about how much pain has interfered with their life, how they have been feeling recently, and thoughts or feelings they have had about their pain problem. These extra questions take about 25 minutes in total to answer.

Subjects will have the option to:

1. complete the extra set of questions all at once, in one of the four telephone interviews,
2. spread the set of questions across the four telephone interviews, so that each call is about 10 minutes long, or
3. complete a bare minimum of questions over the telephone during any of the four phone interviews, and then complete the remaining questions via a paper-and-pencil questionnaire sent to the subject. Subjects will then return the completed questionnaire in a postage-paid envelope provided by staff. Research staff will call subjects if they have not received the completed questionnaire after a certain period of time.

The four telephone interviews must be completed within one week, and each of the assessment calls will take place on different days during the one week. The pre-treatment assessments must be completed in the week before the first treatment session. Otherwise, the first treatment session will be postponed until all four of the assessments have been completed.

Treatment Once subjects are enrolled in the research study and have completed the cognitive testing session and the baseline assessment, a research staff member will call each subject to schedule the initial treatment session. The clinicians who will conduct the treatment sessions are clinical psychologists or trained therapists who are supervised by clinical psychologists.

Before the first treatment session, subjects will be randomly assigned (by chance, like flipping a coin) to one of two treatment interventions. Both treatments involve eight hour-long telephone calls with the assigned study therapist. Both treatments involve educating subjects about pain, discussing the impact of pain, and discussing different ways to manage it in hopes of decreasing subjects' pain and its impact on their lives. Subjects will be encouraged to use what they learn in the telephone sessions outside of treatment to help them with their pain.

Every participant will receive eight 60-minute sessions conducted by telephone by one of the study's clinicians. Whenever possible, research staff will try to schedule the treatment sessions an average of once a week, so that a subject's total time in treatment is eight weeks. Research staff will send subjects a workbook by standard mail or electronically, with materials to refer to and discuss during the telephone sessions, as well as additional materials to review between sessions. Subjects may also receive audio recordings as part of the material they will talk about in treatment.

The research staff members who are conducting the assessments will not know which treatment intervention subjects have been assigned to, nor will they have access to any information covered during the treatment sessions with study clinicians. All treatment is administered over the phone.

Subjects will be asked to complete the follow-up assessments if they decide they no longer want to participate in the study before they finish the treatment sessions.

The study clinician who conducted the treatment sessions will call each subject 2, 6, and 10 weeks after the last treatment session. The clinician will call to ask how subjects are doing and answer questions they may have. These telephone calls are called "booster sessions" and will take about up to 15 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* Veteran Status
* Diagnosis of TBI of any severity verified in VA medical records (e.g., VA TBI Comprehensive Evaluation or other comparable neuropsychological or medical evaluation in the record)
* Most recent TBI must have occurred after onset of OEF
* Military Service in OEF, OIF, and/or OND
* Average pain intensity in the past month of 4 or above on 0-10 numeric rating scale (moderate pain and above)
* Pain of at least six months duration, with pain reportedly present greater than or equal to half of the days in the past six months
* Able to read and speak English
* Able to communicate over the phone (i.e., must be verbal)
* Age 18 years or older

Exclusion Criteria:

* Hospitalization for psychiatric reasons involving psychosis other than suicidal ideation, homicidal ideation, and/or PTSD
* Communication limitations that would prevent ability to participate in the intervention or assessments
* Cognitive impairment that interferes with ability to engage in the intervention despite modifications specifically for TBI. This will be defined as a score of 5/10 or less indicating moderate or severe cognitive impairment on the Short Portable Mental Status Questionnaire (SPMSQ)
* Diagnosis of primary psychotic or major thought disorder as listed in participant's medical record or self-reported

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
average pain intensity in the past week | 10-12 weeks following randomization (post-treatment)
  Average pain intensity will be assessed using an 11-point numerical rating scale (NRS), where 0 means "no pain" and 10 means "pain as bad as you can imagine", accompanied by the following instructions: "Please rate your pain by indicating the number that best describes your pain on average in the last 24 hours".This NRS will be administered by research staff via telephone assessments four times within the week before treatment begins following enrollment into the study and before randomization (pre-treatment), approximately halfway (4 to 6 weeks following randomization) through treatment (mid-treatment), 10-12 weeks following randomization (post-treatment), and 6 months following randomization (6-month). The arithmetic mean of the four ratings at 10-12 weeks following randomization will be used as the primary outcome measure of average pain level.

SECONDARY OUTCOMES:
average pain intensity in the past week | 6 months following randomization
  Average pain intensity will be assessed using an 11-point numerical rating scale (NRS), where 0 means "no pain" and 10 means "pain as bad as you can imagine", accompanied by the following instructions: "Please rate your pain by indicating the number that best describes your pain on average in the last 24 hours".This NRS will be administered by research staff via telephone assessments four times within the week before treatment begins following enrollment into the study and before randomization (pre-treatment), approximately halfway (4 to 6 weeks following randomization) through treatment (mid-treatment), 10-12 weeks following randomization (post-treatment), and 6 months following randomization (6-month). The arithmetic mean of the four ratings at 6 months following randomization will be used as the secondary outcome measure of average pain level to determine whether treatment effects can be maintained over time.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne M Hoffman, PhD, Principal Investigator — University of Washington
Locations (4):
- United States (4):
  - University of Washington, Ninth and Jefferson Building, Seattle, Washington
  - Veteran Affairs Puget Sound Health Care System, Seattle, Seattle, Washington
  - University of Washington, Health Sciences Building, Seattle, Washington
  - VA Puget Sound Health Care System, American Lake, Tacoma, Washington

REFERENCES:
- [Derived] Miller M, Williams R, Pagulayan K, Barber J, Ehde DM, Hoffman J. Correlates of sleep disturbance in Veterans with traumatic brain injury and chronic pain: A cross-sectional study. Disabil Health J. 2022 Jan;15(1):101203. doi: 10.1016/j.dhjo.2021.101203. Epub 2021 Aug 27. PMID 34479850
- [Derived] Hoffman JM, Ehde DM, Dikmen S, Dillworth T, Gertz K, Kincaid C, Lucas S, Temkin N, Sawyer K, Williams R. Telephone-delivered cognitive behavioral therapy for veterans with chronic pain following traumatic brain injury: Rationale and study protocol for a randomized controlled trial study. Contemp Clin Trials. 2019 Jan;76:112-119. doi: 10.1016/j.cct.2018.12.004. Epub 2018 Dec 13. PMID 30553077

DOCUMENTS (1):
  • Informed Consent Form (2016-08-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT01768650/ICF_000.pdf